CLINICAL TRIAL: NCT02489162
Title: The Role of MyotonPro in Assessing the Biomechanical Properties of Facial Muscles in Facial Paralysis Patients and Its Role in Monitoring Recovery Following Facial Reanimation Surgery
Brief Title: The Role of a Device to Evaluate the Neuromuscular Function in Assessing Muscle in Facial Paralysis Patients
Acronym: MyotonPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MiMuMS
Record Dates: First submitted 2015-06-10; First posted 2015-07-02 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2018-10

CONDITIONS: Facial Nerve Palsy
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MyotonPRO (Experimental): Experimental: Measurement of biomechanical properties of mimic muscles on the ipsilateral palsy side with the healthy contralateral side ( case - control design)
  Interventions: Device: MyotonPRO; Device: non-invasive electromyography (EMG)
- Non-invasive electromyography (EMG) (Active Comparator): Comparing experimental intervention with gold standard
  Interventions: Device: MyotonPRO; Device: non-invasive electromyography (EMG)

INTERVENTIONS:
Device: MyotonPRO — MyotonPRO measurements of the biomechanical properties of facial mimic muscles
Device: non-invasive electromyography (EMG) — Gold standard technique for measuring muscle

SUMMARY:
The objective of the research is to determine whether the MyotonPRO has a valid and reliable application in facial, head and neck surgery. In addition, the study aims to compare this new technology with current electromyography.

DETAILED DESCRIPTION:
Facial paralysis has significant aesthetic, functional and psycho-social morbidity. The diagnosis and monitoring of neuromuscular recovery is limited to clinical examination, electromyography (EMG) and electroneurography (ENoG). EMG and ENoG is invasive for the patient and has practical and cost disadvantages. The MyotonPRO is a handheld device, which is pain-free and quick to use. Therefore this research is assessing MyotonPRO technology for this clinical application and may be effective at evaluating rehabilitative and surgical interventions. Phase 1 - Variation of measurements Phase 2 - Mimic muscle dysfunction assessment Phase 3 - Peri-operative Mimic and temporalis muscle assessment Phase 4 - Phase 3 including electromyography Phase 5 - Temporalis and mimic muscle assessment following facial reanimation surgery

ELIGIBILITY:
Inclusion Criteria:

1. unilateral peripheral facial nerve palsy
2. Mental capacity to give consent
3. The patient is able to sit independently

Exclusion Criteria:

1. Adults who have undertaken strenuous exercise within the last twenty-four hours
2. Adults taking prescription medication with a known effect on the mechanical properties of muscle (e.g. benzodiazepines) or receiving antispasmodic medications (e.g. botulinum A toxin)
3. Adults with poor mobility (unable to lie prone).
4. Adults with a body mass index (BMI) >30 kg/m2 . Muscle measurements may be inaccurate with excessive subcutaneous tissue

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Muscle tone (Hz) | 12 months
  Determine the feasibility of the MyotonPRO for assessing biomechanical properties of mimic muscles.

SECONDARY OUTCOMES:
stiffness (N/m) | 12 months
  Determine the feasibility of the MyotonPRO for assessing biomechanical properties of mimic muscles.

OTHER OUTCOMES:
elasticity (Logarithmic decrement) | 12 months
  Determine the feasibility of the MyotonPRO for assessing biomechanical properties of mimic muscles.

CONTACTS AND LOCATIONS:
Overall Officials: John Blythe, FRCS, Principal Investigator — European Face Centre, Universitair Ziekenhuis Brussel and University of Southhampton; Maurice Mommaerts, Prof.Dr.Mult, Study Chair — European Face Centre, Universitair Ziekenhuis Brussel; Daniel Labbé, MD, Study Director — Saint Martin Private Hospital Caen
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No